CLINICAL TRIAL: NCT05021315
Title: Effect of Vaginal Cleaning Using Povidone Iodine Before CS to Reduce Postoperative Wound Infection
Brief Title: Vaginal Cleaning Using Povidone Iodine Before CS to Reduce Postoperative Wound Infection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, ahmed nagy shaker ramadan, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 82019
Record Dates: First submitted 2021-08-20; First posted 2021-08-25 (Actual); Last update posted 2022-07-18 (Actual); Status verified 2022-07

CONDITIONS: Cesarean Section Complications; Vaginal Infection; Postoperative Infection
MeSH Terms: conditions — Vaginitis | interventions — Povidone-Iodine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iodine group (Experimental): 50 women who received preoperative vaginal cleansing with 10% povidone-iodine.
  Interventions: Drug: 10% povidone iodine
- Control group (No Intervention): 50 women who did not receive preoperative vaginal cleansing even with tap water.

INTERVENTIONS:
Drug: 10% povidone iodine — 50 women who received preoperative vaginal cleansing with 10% povidone iodine.
  Other Names: Betadine
  Arms: Iodine group

SUMMARY:
The aim of work to assess the effectiveness of preoperative vaginal cleansing with povidone iodine on reduction of post caesarean section wound infection

Research questions:

Does vaginal cleaning using povidone iodine before cesarean section has effect on reduction of postoperative wound infection??

ELIGIBILITY:
Inclusion Criteria:

* 1. Pregnant women who are 37 weeks gestation or more scheduled for elective cesarean section or those in labor with a limited number of vaginal examinations less than 5 times preoperatively.

  2. Pregnant women who are 37 weeks gestation or more with rupture of membranes but duration less than 24 hours

  3. Women consenting to be included in the study.

Exclusion criteria:

1. Abnormally invasive placenta and placenta previa.
2. Intra-partum fever.
3. Prolonged rupture of membranes more than 24 hours
4. History of exposure to radiation treatment for cancer.
5. History of Gynecological infections (PID).
6. History of abdominal infections, e.g., peritonitis.
7. Debilitating diseases like Diabetes mellitus, Thyroid disorders, Cushing disease, abdominal malignancy.
8. Obesity is defined as pregnant BMI >30 kg/m2.
9. History of wound infection or burst abdomen.
10. History suggestive of massive bleeding during previous cesarean section.
11. allergy to iodine-containing solutions
12. Pregnant women with severe anemia defined as Hb <7 g/dl.
13. Cases with intra-abdominal drain deployment are discarded.
14. Obstructed labor with numerous vaginal examinations.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 800 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-10-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative wound complication | 1 week
  Any sign of infection as redness, hotness and tenderness as well as pyrexia occurance in wound postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa A Sleem, MD, Principal Investigator — Ethical and scientific committee
Locations (2):
- Egypt (2):
  - faculty of medicine - Cairo university, Cairo, Kasr El Ainy
  - faculty of medicine, Kasr el ainy hospital, Cairo university, Cairo